CLINICAL TRIAL: NCT02679430
Title: Prospective Analysis of Prostatic Arterial Embolization
Brief Title: Analysis of Prostatic Arterial Embolization for Benign Prostatic Hyperplasia Using Embosphere Microspheres
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was deferred and never approved by the Maimonides Medical Center IRB.
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/12/VA02
Record Dates: First submitted 2015-10-22; First posted 2016-02-10 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2018-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prostate Arterial Embolization (Other): Intervention: Patients will undergo prostatic artery embolization.
  The purpose of this study is to demonstrate the safety and efficacy of the device, Embosphere Microspheres, in prostatic arterial embolization (PAE). PAE, is now an accepted form of treatment for BPH outside of the United States, however few studies have been performed demonstrating safety and efficacy in the US. Embosphere Microsphere is a device that may be used to reduce blood flow to targeted organs. With this research, we would like to show that Embosphere Microsphere may be used for patients with benign hyperplasia of prostate (BPH to reduce blood flow to the prostate gland. This current study is designed to understand the rate of improved BPH symptoms.
  Interventions: Device: Prostate Arterial Embolization

INTERVENTIONS:
Device: Prostate Arterial Embolization — The purpose of this study is to demonstrate the safety and efficacy of the device, Embosphere Microspheres, in prostatic arterial embolization (PAE). PAE, is now an accepted form of treatment for BPH outside of the United States, however few studies have been performed demonstrating safety and efficacy in the US. Embosphere Microsphere is a device that may be used to reduce blood flow to targeted organs. With this research, we would like to show that Embosphere Microsphere may be used for patients with benign hyperplasia of prostate (BPH to reduce blood flow to the prostate gland. This current study is designed to understand the rate of improved BPH symptoms.

SUMMARY:
Investigators hypothesis that arterial embolization of men with symptomatic BPH, analogous to uterine fibroid embolization for women, is safe and effective.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety and efficacy of the device, Embosphere Microspheres, in prostatic arterial embolization (PAE). PAE, is now an accepted form of treatment for BPH outside of the United States, however few studies have been performed demonstrating safety and efficacy in the US. Embosphere Microsphere is a device that may be used to reduce blood flow to targeted organs. With this research, we would like to show that Embosphere Microsphere may be used for patients with benign hyperplasia of prostate (BPH to reduce blood flow to the prostate gland. This current study is designed to understand the rate of improved BPH symptoms.

Patients with moderate to severe lower urinary tract symptoms resulting from BPH are eligible for this study. Specifically, patients that have been on conservative medical therapy for at least 6 months with no relief of symptoms are being asked to participate in this trial. Patients meeting this criterion would traditionally be considered for more invasive treatment options such as surgery. We believe that PAE is an acceptable alternative to the more invasive treatment options currently the standard of care (available) and therefore we are asking you to participate in this study. We would like to demonstrate that PAE utilizing Embosphere Microsphere will improve their symptoms.

The gold standard of treatment for BPH is transurethral resection of the prostate (TURP). It is very effective but is also an invasive open surgical procedure that carries a high risk of sexual dysfunction and incontinence as side effects of the procedure. It is the goal of this study to demonstrate that these complications are not associated with PAE and that PAE will improve symptoms associated with BPH.

Embosphere Microspheres are small biocompatible plastic spheres that are released inside a vessel under x-ray control. Once inside the vessel, the spheres will block the vessel and decrease blood flow to the tissue supplied by that vessel. Embosphere Microspheres have been cleared by the Food and Drug Administration (FDA) for use in the embolization of blood vessels supplying uterine fibroids and vascular tumors. Additionally, they are approved in the European Union for treatment of BPH. This study has been approved by the FDA to use Embosphere Microspheres for research purposes in the treatment of BPH.

ELIGIBILITY:
Inclusion Criteria:

1. Males with the clinical diagnosis of BPH.
2. IPSS >18 with symptoms that are refractory to medical treatment with combination therapy (alpha-blocker + 5-alpha-reductase-inhibitor (5-ARI), as tolerated by the patient) for a minimum of six months.
3. Candidates for Transurethral resection of the prostate (TURP), open prostatectomy, Transurethral Needle Ablation (TUNA), or other procedures such as thermal ablation.
4. Patients are candidates for above procedures, however comorbid conditions present a prohibitive surgical risk.

Exclusion Criteria:

1. Urethral strictures, bladder neck contracture, or other potentially confounding bladder pathology.
2. Neurogenic bladder and/or sphincter abnormalities due to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes, etc.
3. Uncontrolled diabetes mellitus, significant respiratory disease, or known immunosuppression
4. Severe allergy to iodine contrast and unable to be pre-medicated.
5. Allergy to gelatin containing products.
6. Patient is on anticoagulation or anti-platelet treatment and cannot halt medication for 5 days prior to PAE.
7. Patient is unable to have a MRI/MRA performed.
8. Magnetic Resonance Angiogram (MRA) reveals severe aorto-iliac atherosclerotic disease prohibiting intervention.
9. Compromised renal function determined as serum creatinine level > 1.8 mg/dl, or upper-tract disease.
10. Prior diagnosis of any pelvic malignancy including prostate cancer.
11. Have received prior radiation to the pelvis for any condition.
12. Have had prior pelvic surgery or non-medical BPH treatment.

Ages: 35 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Estimated); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 12 months
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  The questions refer to the following urinary symptoms:
  Questions Symptom
  1. Incomplete emptying
  2. Frequency
  3. Intermittency
  4. Urgency
  5. Weak Stream
  6. Straining
  7. Nocturia Question eight refers to the patient's perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Sobolevsky, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No